CLINICAL TRIAL: NCT01990820
Title: A Randomized Trial of the Management of Pediatric Chronic Rhinosinusitis With or Without Balloon Sinusplasty
Brief Title: Study for the Management of Pediatric Chronic Rhinosinusitis With or Without Balloon Sinuplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endeavor Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EH09-177
Record Dates: First submitted 2013-11-16; First posted 2013-11-21 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Rhinitis + Sinusitis, Pediatric Chronic Rhinosinusitis
Keywords: Pediatric Chronic Rhinosinusitis
MeSH Terms: conditions — Rhinitis; Sinusitis | interventions — Adenoidectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adenoidectomy without balloon dilation (Active Comparator): Subjects will have Adenoidectomy + maxillary sinus irrigation, without balloon dilation.
  Interventions: Procedure: Adenoidectomy + Maxillary Sinus Irrigation
- Adenoidectomy with balloon dilation (Experimental): Adenoidectomy + balloon dilation of maxillary sinus ostia using Acclarent Relieva Balloon Sinuplasty + irrigation
  Interventions: Device: Acclarent Relieva Balloon Sinuplasty

INTERVENTIONS:
Device: Acclarent Relieva Balloon Sinuplasty — A rigid nasal endoscopy will be performed. After decongesting with oxymetazoline hydrochloride, the balloon catheter device will be inserted and the wire/balloon will be threaded through the maxillary sinus ostia. Confirmation of location will be per manufacturer's recommendation with either fluoroscopy or illumination. Following confirmation, the balloon will be dilated under visualization per manufacture's recommendation. After the visualization of the dilated ostia, cultures for aerobic/anerobic examination will be taken and irrigation with 10ml of isotonic sodium chloride will be performed.
  Adenoidectomy will be performed using either the microdebrider or suction electrocautery in the usual manner.
  Other Names: Relieva Sinus Balloon Catheter 510K: K073041; Luma Illumination System 510K: K071845; Guide Cathetheter 510K: K043445; Votex Irrigation Catheter 510K: K043445; Guidewire 510K: K043445; Sidekick 510K: K043445; Inflation Devie 510K: K052198
  Arms: Adenoidectomy with balloon dilation
Procedure: Adenoidectomy + Maxillary Sinus Irrigation — A rigid nasal endoscopy will be performed. After decongesting with oxymetazoline hydrochloride, the maxillary sinuses will be entered via middle meati punctures using either a sterile spinal needle or a curved suction. Sinus contents will be aspirated and sent for aerobic/anaerobic cultures. Irrigation with 10ml of isotonic sodium chloride will be performed. If no material is aspirated initially, the sinus contents will be re-aspirated after irrigation and sent for aerobic/anaerobic cultures.
  Adenoidectomy will be performed using either the microdebrider or suction electrocautery in the usual manner.
  After adequate hemostasis, the patient will be awakened and brought to the recovery room. Depending on the recovery, the child will either be admitted or discharged home.
  Arms: Adenoidectomy without balloon dilation

SUMMARY:
Chronic rhinosinusitis, a common diagnosis in children, remains a poorly understood disease. Adenoidectomy (surgery to take out the adenoid pads- infection fighting glands in the back of the throat) is performed since the adenoid pad may trap germs that enter a child's body and can get so swollen with bacteria that they become infected themselves. Functional endoscopic sinus surgery (FESS) and adenoidectomy are currently the most common surgeries performed on children with this disease. Another treatment is adenoidectomy and irrigation of the maxillary sinus without FESS. New technology has emerged using a balloon catheter to dilate (open) the sinus passage in addition to the adenoidectomy and irrigation. This study seeks to answer if children with chronic rhinosinusitis who undergo adenoidectomy with balloon dilation of the maxillary sinus passage and irrigation experience improved quality of life outcomes compared to children with chronic rhinosinusitis who undergo an adenoidectomy with maxillary sinus irrigation without dilation of the sinus passage.

ELIGIBILITY:
Inclusion Criteria:

1. Sinonasal symptoms of at least 12 weeks' duration or recurrent sinusitis >3x/year
2. Failure to respond to 3-week course of antibiotic and 3 month course of nasal steroid preparations or antihistamines as well as saline nasal irrigation
3. Rhinosinusitis documented by CT scan following oral antibiotic course.

Computer tomographic findings considered to be consistent with sinusitis include partial or complete sinus opacification.

Allergy and immunology workup will be recommended on an individual basis -

Exclusion Criteria:

1. Patients with extensive sinonasal polyps, extensive sinonasal osteoneogenesis, sinonasal tumors
2. History of facial trauma that distorts sinus anatomy
3. Ciliary dysfunction
4. Pregnancy will be excluded.
5. Patients with cystic fibrosis, craniofacial anomalies, metabolic disorders, or immunodeficiencies
6. Patients who have had their adenoids removed and thus may be candidates for functional endoscopic sinus surgery will also be excluded.
7. Patients with a history of sinus surgery or significant anatomic abnormalities on CT scan that would require endoscopic sinus surgery or septoplasty would also be excluded.

Of note, children who will be undergoing concurrent surgeries will not be excluded.

-

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2009-03; Primary Completion 2016-09-29 (Actual); Study Completion 2016-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Gerber, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 4 participants were enrolled on incorrect consent forms so their data were not collected. The IRB provided approval to enroll additional patients to make up for these 4 patients.
Groups:
- Arm 1: Subjects will have Adenoidectomy + maxillary sinus irrigation, without balloon dilation.
  Adenoidectomy + Maxillary Sinus Irrigation: A rigid nasal endoscopy will be performed. After decongesting with oxymetazoline hydrochloride, the maxillary sinuses will be entered via middle meati punctures using either a sterile spinal needle or a curved suction. Sinus contents will be aspirated and sent for aerobic/anaerobic cultures. Irrigation with 10ml of isotonic sodium chloride will be performed. If no material is aspirated initially, the sinus contents will be re-aspirated after irrigation and sent for aerobic/anaerobic cultures.
  Adenoidectomy will be performed using either the microdebrider or suction electrocautery in the usual manner.
  After adequate hemostasis, the patient will be awakened and brought to the recovery room. Depending on the recovery, the child will either be admitted or discharged home.
- Arm 2: Adenoidectomy + balloon dilation of maxillary sinus ostia using Acclarent Relieva Balloon Sinuplasty + irrigation
  Acclarent Relieva Balloon Sinuplasty: A rigid nasal endoscopy will be performed. After decongesting with oxymetazoline hydrochloride, the balloon catheter device will be inserted and the wire/balloon will be threaded through the maxillary sinus ostia. Confirmation of location will be per manufacturer's recommendation with either fluoroscopy or illumination. Following confirmation, the balloon will be dilated under visualization per manufacture's recommendation. After the visualization of the dilated ostia, cultures for aerobic/anerobic examination will be taken and irrigation with 10ml of isotonic sodium chloride will be performed.
  Adenoidectomy will be performed using either the microdebrider or suction electrocautery in the usual manner.
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.0 (2.9) | 6.5 (2.1) | 6.75 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 6 | 6 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life (QoL) Outcomes Between Adenoidectomy + Maxillary Sinus Irrigation With or Without the Use of Balloon Dilation or Maxillary Sinus Ostia.
Description: The care giver for each subject will be asked to complete SN-5 Pediatric sinonasal symptom survey (SN-5) at baseline (prior to surgery) and 6 and 12 months post surgery.
  The SN-5 is a health-related qualify of life (QOL) questionnaire which consists of 5 questions about sinus problems (sinus infection, nasal obstruction, allergy symptoms, emotional distress, activity limitations) each of which is scored by the caregiver on a 7 point response scale. The 5 responses are then averaged into an SN-5 overall score (1-7). 1 is the minimum value for the overall SN-5 (best QoL) and 7 is the maximum value (worst QoL) The questionnaire also asks the caregiver to grade overall health related quality of life using a visual analog scale from 0 (worse possible quality of life) to 10 (best possible quality of life). The visual analog scale is scored separately from the SN-5 average score.
Time Frame: 6 and 12 months postoperatively
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adenoidectomy Without Balloon Dilation | Adenoidectomy With Balloon Dilation
Number analyzed (Participants) | 13 | 12
score on a scale
  SN-5 overall score (6 months postoperatively) | 2.48 (0.62) | 2.5 (1.42)
  SN-5 overall score (12 months postoperatively | 2.25 (0.86) | 2.40 (1.11)
  Quality of Life score (6 month) | 8.10 (0.88) | 8.27 (2.10)
  Quality of Life score (12 months) | 8.27 (1.27) | 7.60 (1.71)

ADVERSE EVENTS:
Groups:
- Arm 1: Subjects will have Adenoidectomy + maxillary sinus irrigation, without balloon dilation.
- Arm 2: Adenoidectomy + balloon dilation of maxillary sinus ostia using Acclarent Relieva Balloon Sinuplasty + irrigation
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 0/13 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No